CLINICAL TRIAL: NCT00008268
Title: A Phase II Study Of Blood Stem Cell Mobilization With Intravenous Melphalan (60 MG/M2) + G-CSF In Patients With Multiple Myeloma
Brief Title: Melphalan and Filgrastim to Stimulate Peripheral Stem Cells in Patients With Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 00-067; CDR0000068392 (Registry Identifier: PDQ (Physician Data Query)); NCI-G00-1895
Record Dates: First submitted 2001-01-06; First posted 2003-01-27 (Estimated); Last update posted 2013-06-18 (Estimated); Status verified 2013-06

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Filgrastim; Melphalan

INTERVENTIONS:
Biological: filgrastim
Drug: melphalan

SUMMARY:
RATIONALE: Melphalan and colony-stimulating factors such as filgrastim may increase the number of immune cells found in bone marrow or peripheral blood.

PURPOSE: Phase II trial to study the effectiveness of melphalan combined with filgrastim in stimulating peripheral stem cells in patients who have multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety and efficacy of melphalan when used with filgrastim (G-CSF) for stem cell mobilization in patients with multiple myeloma.
* Analyze how this mobilization regimen affects parameters of stem cell (CD34+) mobilization and collection in these patients.
* Determine how this mobilization regimen affects disease status and clonotypic (i.e., tumor cell) contamination in stem cell components in these patients.

OUTLINE: Patients undergo peripheral blood stem cell (PBSC) mobilization consisting of melphalan IV on day 1 and filgrastim (G-CSF) subcutaneously beginning on day 2 and continuing until PBSC collection is complete.

Patients are followed at 1 month.

PROJECTED ACCRUAL: A total of 11-32 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of multiple myeloma
* Must have received induction therapy within the past 3 months
* Chemoresponsive disease

  * Greater than 50% reduction of monoclonal paraprotein with reduction in marrow plasma cell infiltrate or greater than 50% reduction in marrow plasma cell infiltrate if disease is non-secretory
* No symptomatic pleural effusions
* Eligible for stem cell transplantation

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-3 (ECOG 3 allowed only if due to bone disease or neuropathy)

Life expectancy:

* Not specified

Hematopoietic:

* Platelet count at least 150,000/mm^3

Hepatic:

* Bilirubin no greater than 2.5 mg/dL

Renal:

* Creatinine no greater than 2.5 mg/dL OR
* Creatinine clearance greater than 51 mL/min

Cardiovascular:

* No symptomatic cardiomyopathy
* No medically documented symptomatic cardiac arrhythmias within the past 60 days
* No New York Heart Association class III congestive heart failure
* No myocardial infarction within the past 6 months

Other:

* No other concurrent medical conditions that would preclude study
* No uncontrolled infections
* No other active malignancy within the past 5 years except for non-melanoma skin cancer
* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior stem cell mobilization or transplantation

Chemotherapy:

* See Disease Characteristics
* No more than 200 mg prior oral melphalan

Endocrine therapy:

* Not specified

Radiotherapy:

* No more than 3000 cGy of prior radiotherapy for myeloma

Surgery:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-08; Primary Completion 2003-06 (Actual); Study Completion 2003-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raymond L. Comenzo, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States